CLINICAL TRIAL: NCT07135271
Title: Building and Evaluating a Stratified Prostate Cancer Pathway (BeSpoke): the Impact of BeSpoke Decision Support in Patients With Newly Diagnosed Localised Prostate Cancer - a Single-blind Randomised Controlled Trial With Mixed Method Analysis
Brief Title: BeSpoke Decision Support for Patients With Newly Diagnosed Localised Prostate Cancer
Acronym: BeSpoke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 176848; IRAS 347220 (Other: NHS Health Research Authority); 25/LO/0394 (Other: London - Fulham Research Ethics Committee)
Record Dates: First submitted 2025-08-11; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Localised Prostate Cancer
Keywords: Localised Prostate Cancer; Patient Decision Aid; Shared Decision Making; Randomised Clinical Trial
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Placebo Comparator): Standard of Care Counselling information
  Interventions: Other: Standard of Care (SOC) decision support material
- BeSpoke Decision Support (Experimental): Standard of care counselling plus access to BeSpoke Decision Support tool
  Interventions: Other: Bespoke Decision Support tool; Other: Standard of Care (SOC) decision support material

INTERVENTIONS:
Other: Bespoke Decision Support tool — A newly-developed online patient decision aid offering comparative information of prostate cancer treatments (active surveillance, focal therapy, radical prostatectomy and external beam radiotherapy), personalised estimates of oncological and functional outcomes for each treatment and a value-clarification exercise.
  Arms: BeSpoke Decision Support
Other: Standard of Care (SOC) decision support material — Standard of care information to inform the prostate cancer treatment decision. This includes the nationally approved Prostate Cancer UK information booklet "Prostate Cancer - A guide if you have just been diagnosed" in all sites. Further educational material may be provided as part of standard of care depending on local practice at each site.

SUMMARY:
The goal of this randomised clinical trial is to assess whether personalised treatment counselling can improve the decision-making experience in patients with a new diagnosis of localised prostate cancer. The main question it aims to answer is:

• Does the Bespoke Decision Support tool reduce decisional conflict in those choosing between treatment options for localised prostate cancer?

Researchers will compare the addition of the Bespoke Decision Support tool to standard treatment counselling versus standard counselling alone.

Patient participants will:

* Receive standard counselling with or without access to the Bespoke Decision Support tool (based on arm of randomisation), prior to making a treatment decision.
* Answer to questionnaires regarding urinary, sexual and bowel function and decision-making outcomes before and after making a treatment decision and at 3, 6, and 12 months after initiating treatment.
* Take part in a qualitative interview to discuss their decision-making experience

Health Care Professional participants will:

• Take part in a qualitative interview to discuss their experience in providing decision support in the trial using the Bespoke Decision Support tool.

DETAILED DESCRIPTION:
Recruited patient participants will be randomised into two arms:

* Standard of Care (SOC) arm: SOC counselling
* Intervention arm: SOC counselling plus access to BeSpoke Decision Support

The standard of care (SOC) arm includes the nationally-approved Prostate Cancer UK booklet "Prostate Cancer - A guide if you have recently been diagnosed" and patient appointments to discuss different treatments with clinicians, as per local practice that offer them. Further educational material may be provided as per local practice at each site.

The intervention arm will offer additional BeSpoke Decision Support providing:

* Consistent and up-to-date information about suitable treatment approaches.
* Risk-stratified predictions of treatment outcomes based on baseline cancer and patient characteristics.
* Value clarification about which attributes of treatment are most important to the individual.

All participants will complete questionnaires on demographic data, functional status and measures of decision-making experiences at several time points: enrolment (prior to treatment discussion consultation); after treatment decision has taken place; at 3, 6, and 12 months after treatment commences.

The investigators will interview health care professionals and a sample of patient participants to assess the effect of the BeSpoke Decision Support and the challenges in implementation across the NHS.

ELIGIBILITY:
Inclusion Criteria for Patient-Participants:

1. Newly diagnosed localised prostate cancer
2. Clinically suitable for at least two of the following treatment options:

   1. active surveillance
   2. focal therapy
   3. radical prostatectomy
   4. external beam radiotherapy
3. Willing and able to provide informed consent

Exclusion Criteria for Patient Participants:

1. Unsuitable for active treatment due to very low risk prostate cancer or significant health issues.
2. Suspicion of metastatic prostate cancer based on clinical or imaging evidence including:

   1. Imaging identified suspicious lesion on bone scan, CT, whole-body MRI or PSMA-PET/CT;
   2. PSA ≥50 ng/mL.
3. Not able to provide informed consent.
4. Insufficient English proficiency for adequate use of BeSpoke Decision Support. (Patients with support from a family member, friend or partner, to overcome lack of English proficiency will be included.)
5. Enrolled in other localised prostate cancer studies where treatment is assigned rather than chosen by participants, e.g. PART Trial (Partial prostate Ablation vs Radical prostaTectomy)

Inclusion criteria for Health Care Professionals:

1. Have seen BeSpoke Decision Support and spoken to patients in the intervention arm.
2. Willing and able to provide written or electronic informed consent

Exclusion criteria for Health Care Professionals

1. No experience of BeSpoke Decision Support.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) | After treatment decision is confirmed, assessed as patient-reported outcome measure via questionnaire delivered on average after 4 weeks from enrolment.
  Mean difference in DCS between control (SOC) arm and intervention (Bespoke Decision Support) groups.
  Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].

SECONDARY OUTCOMES:
Preparation for Decision Making (PrepDM) Scale | After treatment decision is confirmed, assessed as patient-reported outcome measure via questionnaire delivered on average after 4 weeks from enrolment.
  Mean difference in PrepDM Scale between control and intervention group. Scores range from 0 to 100 [higher scores indicate higher perceived level of preparation for decision making].
Decision Self Efficacy (DSE) Scale | After treatment decision is confirmed, assessed as patient-reported outcome measure via questionnaire delivered on average after 4 weeks from enrolment.
  Mean difference in the DSE score between the control and the intervention groups.
  Scores range from 0 [not at all confident] to 100 [very confident].
Satisfaction With Decision (SWD) Scale | Measured at multiple time points: after treatment decision is confirmed (assessed as patient-reported outcome measure via questionnaire delivered on average after 4 weeks from enrolment); and at 3, 6 and 12 months from the treatment date.
  Mean difference in the SWD score between the control and the intervention groups. Scores range from 1 to 5 (5=higher satisfaction).
Decision Regret Scale (DRS) | Measured at multiple time points: after treatment decision is confirmed (assessed as patient-reported outcome measure via questionnaire delivered on average after 4 weeks from enrolment); and at 3, 6 and 12 months from the treatment date.
  Mean difference in the DRS score between the control and the intervention groups.
  Scores range from 0 [no regret] to 100 [high regret].
Satisfaction with Cancer Information Profile (SCIP) Scale | Measured after treatment decision is confirmed (assessed as patient-reported outcome measure via questionnaire delivered on average after 4 weeks from enrolment) and at 12 months after treatment initiation.
  Mean difference in the SCIP score between the control and the intervention groups at time-point 1 and time-point 4.
  Scores for the sub-scale "Satisfaction with the amount and content of information" range from 1 to 14 (14=higher satisfaction).
  Scores for the sub-scale "Satisfaction with the form and timing of information" range from 7 (lower satisfaction) to 35 (higher satisfaction).
Control Preference Scale (CPS) | Measured at enrolment and after treatment decision is confirmed (assessed as patient-reported outcome measure via questionnaire delivered on average after 4 weeks from enrolment).
  Frequencies and proportion of the CPS categories in both the intervention and the control group.
Hospital Anxiety and Depression Scale (HADS) | Measured before giving intervention, and after 3, 6 and 12 months from treatment initiation.
  Frequencies and proportion of the HADS categories in both the intervention and the control group.
  Scores range from 0 to 21: 0-7 = Normal; 8-10 = Borderline abnormal (borderline case); 11-21 = Abnormal (case).
Decisional Conflict Scale (DCS) Subscales | After treatment decision is confirmed, assessed as patient-reported outcome measure via questionnaire delivered on average after 4 weeks from enrolment.
  Means or medians of the intervention and the control groups for the different DCS sub-scores:
  * Informed sub-score (Scores range from 0 [feels extremely informed] to 100 [feels extremely uninformed]);
  * Values Clarity sub-score(Scores range from 0 [feels extremely clear about personal values for benefits & risk/side effects] to 100 [feels extremely unclear about personal values]);
  * Support sub-score (Scores range from 0 [ feels extremely supported in decision making] to 100 [feels extremely unsupported in decision making]);
  * Uncertainty sub-score (Scores range from 0 [feels extremely certain about best choice] to 100 [feels extremely uncertain about best choice]);
  * Effective Decision sub-score (Scores range from 0 [good decision] to 100 [bad decision]).
Qualitative Assessment with Patients | Between treatment decision being recorded and end of study (12 months after treatment initiation)
  Qualitative interview evaluating patient experience in treatment decision making and feedback on decision support material
Qualitative assessment with Health Care Professionals (HCP) | Through study completion, an average of 1 year
  Qualitative interviews with HCP (urologists, clinical oncologists, clinical nurse specialists, GPs) involved in the treatment decision making pathway of patients with prostate cancer, to inquire regarding the decision support material provided as standard of care and in the intervention arm.

OTHER OUTCOMES:
Number of treatment counselling consultations | From date of randomisation until the date of first documented recording of treatment decision, assessed up to 12 months.
  Mean or median difference in number of treatment counselling consultations taking place between enrolment and treatment decision between the control and intervention group.
Treatment choice | From date of randomisation until the date of first documented recording of treatment decision, assessed up to 12 months.
  Proportion of different treatments chosen (active surveillance, focal therapy, radical prostatectomy and radiotherapy) between the intervention and the control groups.
Time to treatment decision | From date of randomisation until the date of first documented recording of treatment decision, assessed up to 12 months.
  Time passed between enrolment and recording of treatment decision between the control and intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Moore, MD, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: No
Any request to share IPD from other researchers will be evaluated by the Trial Steering Committee on an ad hoc basis.

REFERENCES:
- See also: Prostate Cancer: A guide if you've just been diagnosed - Prostate Cancer UK — https://shop.prostatecanceruk.org/pdf/publication/prostate-cancer-a-guide-if-youve-just-been-diagnosed_ifm.pdf